CLINICAL TRIAL: NCT05968833
Title: Addressing the Mental Health Needs of Parents of Pediatric Kidney Transplant Recipients With the iParent2Parent Peer Support Program
Brief Title: iParent2Parent Peer Support Program for Parents of Pediatric Kidney Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Samantha Anthony, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000080780
Record Dates: First submitted 2023-06-29; First posted 2023-08-01 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Kidney Transplant
Keywords: Peer Support Mentorship; Parent Support Mentorship; Pediatrics; Transplant

STUDY DESIGN:
Intervention Model Description: Pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iParent2Parent Program (Experimental)
  Interventions: Behavioral: iParent2Parent Program

INTERVENTIONS:
Behavioral: iParent2Parent Program — iParent2Parent is an online peer support mentorship program that is based on the iPeer2Peer online peer support mentorship program, which has been established in multiple chronic disease populations as a self-management intervention, including in chronic pain and juvenile idiopathic arthritis populations. The iParent2Parent program connect parents one-to-one with other parents of pediatric kidney transplant recipients who are trained to offer vital peer support and mentorship.

SUMMARY:
The iParent2Parent (iP2P) program is a new, innovative virtual mentorship program that will connect parents one-to-one with other parents of pediatric kidney transplant recipients who are trained to offer vital peer support and mentorship. Parents of children who received a kidney transplant at The Hospital for Sick Children will be invited to participate as mentors and mentees. The iP2P program can decrease feelings of isolation, improve mental health and have a long-term positive impact on patient health. This research will increase our understanding of one-to-one peer support and leverage eHealth technologies to improve the access to and acceptability of parent peer support interventions.

ELIGIBILITY:
Mentee Inclusion Criteria:

* Parent of a patient under 18 years of age who received a kidney transplant and is at least two months post-transplant,
* Access to a device (e.g., smart phone, tablet, computer) capable of using free WhatsApp software, and
* English-speaking.

Mentor Inclusion Criteria:

* Parent of a patient under 21 years of age who received a kidney transplant and is at least one year post-transplant,
* Nominated by their child's healthcare team as a good candidate to act in the mentor role (e.g., good communication skills, positive adaptation and adjustment post-transplant, strong support network),
* Access to a device (e.g., smart phone, tablet, computer) capable of using free WhatsApp software, and
* English-speaking.

Exclusion Criteria:

* Non-English speaking.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates and withdrawal rates | Baseline to study completion, an average of 1 year
  How many participants were recruited and have withdrawn from the program on average.
Adherence with the iParent2Parent program | Baseline to study completion, an average of 1 year
  When the participant completes 10 audio or video calls over 12 weeks and 100% when all online outcome measures completed.
Acceptability (Mentees) | Baseline to 12 weeks after baseline/immediately after the intervention
  Whether the innovation is agreeable, palatable or satisfactory.
  Measured via semi-structured interview or focus group.
Acceptability (Mentors) | Baseline to program completion, an average of one year
  Whether the innovation is agreeable, palatable or satisfactory.
  Measured via semi-structured interview or focus group.
Level of engagement with the iParent2Parent program (Mentees) | Baseline to 12 weeks after baseline/immediately after the intervention
  Measured via semi-structured interview or focus group.
Level of engagement with the iParent2Parent program (Mentors) | Baseline to program completion, an average of one year
  Measured via semi-structured interview or focus group.
Barriers and enablers of the iParent2Parent program (Mentees) | Baseline to 12 weeks after baseline/immediately after the intervention
  Measured via semi-structured interview or focus group.
Barriers and enablers of the iParent2Parent program (Mentors) | Baseline to program completion, an average of one year
  Measured via semi-structured interview or focus group.

SECONDARY OUTCOMES:
Parenting stress (Mentees and Mentors) | Baseline to program completion, an average of one year
  Parental Stress Scale; 18-item questionnaire. Each question is scored on a scale from 1 to 5, with scores ranging from 18 to 90. An overall higher score means a worse outcome.
Psychological distress (Mentees and Mentors) | Baseline to program completion, an average of one year
  General Anxiety Disorder-7; 7-item questionnaire. Each question is scored on a scale from 0 to 3, with scores ranging from 0 to 21. An overall higher score means a worse outcome.
Psychological distress (Mentees and Mentors) | Baseline to program completion, an average of one year
  Patient Health Questionnaire Depression Scale; 8-item questionnaire. Each question is scored on a scale from 0 to 3, with scores ranging from 0 to 24. An overall higher score means a worse outcome.
Perceived social support (Mentees and Mentors) | Baseline to program completion, an average of one year
  Short form version 2.0 of the PROMIS battery for: Social Isolation; 6-item questionnaire. Each question is scored on a scale from 1 to 5 and generates a T-score. An overall higher score means a worse outcome.
Perceived social support (Mentees and Mentors) | Baseline to program completion, an average of one year
  Short form version 2.0 of the PROMIS battery for: Informational Support; 6-item questionnaire. Each question is scored on a scale from 1 to 5 and generates a T-score. An overall higher score means a better outcome.
Perceived social support (Mentees and Mentors) | Baseline to program completion, an average of one year
  Short form version 2.0 of the PROMIS battery for: Emotional Support; 6-item questionnaire. Each question is scored on a scale from 1 to 5 and generates a T-score. An overall higher score means a better outcome.
Coping (Mentees and Mentors) | Baseline to program completion, an average of one year
  Coping Health Inventory for Parents; 16-item questionnaire. Each question about coping behaviour is scored on a scale from 0 to 3, with a possible response of "Did not use" the coping behaviour. Scores range from 0 to 48. An overall higher score means a better outcome.
Family Functioning (Mentees and Mentors) | Baseline to program completion, an average of one year
  Pediatric Quality of Life Inventory(TM) 2.0 Family Impact Module; 36-item questionnaire with 8 different sections: Physical Functioning, Emotional Functioning, Social Functioning, Cognitive Functioning, Communication, Worry, Daily Activities, and Family Relationships. Each question is scored on a scale from 0 to 4. Items are reverse-scored and linearly transformed to a 0-100 scale. An overall higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha J. Anthony, PhD, MSW, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No